CLINICAL TRIAL: NCT05748964
Title: Different Surgical Approaches for Treatment of UPJ Obstruction in Children: Prospective Randomized Clinical Trial
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Kamel Ali Mohamed, Mr., Assiut University
Other Study IDs: AKA1712
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Urologic Diseases; Surgery
Keywords: UPJ obstruction; pediatric urology; pyeloplasty
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transperitoneal approach laparoscopic pyeloplasty. (TALP): Transperitoneal approach laparoscopic pyeloplasty. (TALP)
  Interventions: Procedure: Laparoscopic pyeloplasty
- Retroperitoneal Approach laparoscopic pyeloplasty. (RALP): Retroperitoneal Approach laparoscopic pyeloplasty. (RALP)
  Interventions: Procedure: Laparoscopic pyeloplasty

INTERVENTIONS:
Procedure: Laparoscopic pyeloplasty — Twenty patients presented with ureteropelvic junction obstruction [UPJO] will be divided into two equal groups. The first was subjected to trans-peritoneal pyeloplasty while the second was subjected to retroperitoneal pyeloplasty.

SUMMARY:
This study aimed to evaluate the clinical efficacy of laparoscopic pyeloplasty (LP) for ureteropelvic junction obstruction (UPJO) via retroperitoneal and transperitoneal approaches.

DETAILED DESCRIPTION:
Ureteropelvic junction obstruction (UPJO) is the most common congenital abnormality of the kidney and is responsible for flank pain, recurrent urinary infections, hydronephrosis and the loss of renal function. Until recently, open pyeloplasty (OP) was the standard surgical treatment modality for UPJO.However, with the development of laparoscopic devices and surgical technology, laparoscopic pyeloplasty (LP) has become a more beneficial choice for the patients with UPJO than open surgery because of the advantages of excellent visualization, minimal trauma, rapid postoperative recovery, good cosmetic result, and a nearly successful rate compared with open pyeloplasty. The first LP in children was performed in 1995. It has gained popularity for older children. LP can be performed though retroperitoneal and transperitoneal approaches. Which surgical method is better is still controversial.

ELIGIBILITY:
Inclusion Criteria:

* Age above two years.
* Unilateral UPJO.

Exclusion Criteria:

* Age below two years.
* Bilateral UPJO.
* Recurrent UPJO.
* Malrotated kidneys and renal fusion anomalies.

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children diagnosed with unilateral ureteropelvic junction obstruction
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Operative time | From April 1, 2023 to April 1, 2024
  Operative time

SECONDARY OUTCOMES:
Convergence rate | From April 1, 2023 to April 1, 2024
  Convergence to open pyeloplasty
Post operative complications | From April 1, 2023 to April 1, 2024
  Post operative complications
Hospital stay | From April 1, 2023 to April 1, 2024
  Hospital stay

IPD SHARING:
Plan to Share IPD: No